CLINICAL TRIAL: NCT05524493
Title: High-field MR Imaging in Migraine, Visual Snow and Epilepsy
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00936
Record Dates: First submitted 2022-08-18; First posted 2022-09-01 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Migraine; Epilepsy; Visual Snow Syndrome
MeSH Terms: conditions — Migraine Disorders; Epilepsy; visual snow syndrome | interventions — Diffusion Magnetic Resonance Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy participants
  Interventions: Diagnostic Test: Structural MRI; Diagnostic Test: Quantitative MRI; Diagnostic Test: Diffusion MRI; Diagnostic Test: fMRI; Diagnostic Test: MR Spectroscopy
- Patients with migraine
  Interventions: Diagnostic Test: Structural MRI; Diagnostic Test: Quantitative MRI; Diagnostic Test: Diffusion MRI; Diagnostic Test: fMRI; Diagnostic Test: MR Spectroscopy
- Patients with drug resistent epilepsy
  Interventions: Diagnostic Test: Structural MRI; Diagnostic Test: Quantitative MRI; Diagnostic Test: Diffusion MRI; Diagnostic Test: fMRI; Diagnostic Test: MR Spectroscopy
- Patients with visual snow syndrome
  Interventions: Diagnostic Test: Structural MRI; Diagnostic Test: Quantitative MRI; Diagnostic Test: Diffusion MRI; Diagnostic Test: fMRI; Diagnostic Test: MR Spectroscopy

INTERVENTIONS:
Diagnostic Test: Structural MRI — We will examine migraine and epilepsy patients as well as healthy controls using conventional structural MRI in the brain and spinal cord including T1-, T2-, and T2*-weighted sequences
Diagnostic Test: Quantitative MRI — We will examine migraine and epilepsy patients as well as healthy controls using quantitative MRI in the brain and spinal cord. This includes multi-parameter mapping (MPM) and quantitative susceptibility mapping (QSM).
Diagnostic Test: Diffusion MRI — We will examine migraine and epilepsy patients as well as healthy controls using diffusion MRI in both brain and spinal cord.
Diagnostic Test: fMRI — We will examine migraine and epilepsy patients as well as healthy controls using resting-state and task fMRI (including sensory stimulation using pain stimulus) in both brain and spinal cord.
Diagnostic Test: MR Spectroscopy — We will examine migraine and epilepsy patients as well as healthy controls using MR Spectroscopy in both brain and spinal cord.

SUMMARY:
In this project, the aim is to recruit patients with drug resistant epilepsy and those suffering from migraine. Interestingly, patients suffering from epilepsy are also more often reporting to suffer from migraine. The pathobiology is understudied, but it is believed that both etiologies results from brain networks changes. A clinical certified 7T Terra Siemens scanner will be employed to assess in all participants (including healthy controls) how the microstructure differs in disease specific areas. Patients will further be clinically assessed as well as undergo questionnaires.

Migraine is also a common comorbidity to visual snow syndrom and has been shown to impact similar brain regions. However, the pathophysiology is still understudied and a better understanding of the two diseases is needed.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patient must be able to read and sign the informed consent form
* Stable prophylactic medication for 2 months prior to MRI
* At leat one of the two criteria applies:
* Patients diagnosed with migraine (with or without aura, episodic or chronic). Diagnosis is ensured by clinical interview (at least 8 weeks prior to MRI). Also, patients complete a migraine questionnaire (HARDSHIP) (at least 8 weeks before MRI). Migraine frequency ≥ 2 migraine attacks/month.
* Patients with drug resistent epilepsy accroding to ILAE crtieria
* Patients with diagnoses of Visual snow syndrome

Healthy participants;

* No migraine (validated by questionnaire) or epilepsy
* Participants must be able to read and sign the informed consent form

Exclusion Criteria:

* Treatment of migraine disease with Botox within < 4 months before baseline and during the study period
* Pregnant or breastfeeding women
* Intention during the course of the trial to become pregnant
* Women with bilateral ovariectomy, with or without hysterectomy, and postmenopausal women (>2 years of age) are not considered childbearing.
* Other clinically significant comorbidities (e.g., renal insufficiency, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected noncompliance with the protocol, drug or alcohol abuse,
* Patient's inability to follow trial procedures, e.g., due to language problems, mental illness, dementia, etc.,
* Prior participation in the clinical trial
* Enrolment of the investigator, his/ her family members, employees and other dependent persons of the test personnel
* Metallic objects in the body (e.g., splinters, MR incompatible implants).
* Pacemaker
* Claustrophobia
* Obesity (body mass index > 35 kg/m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the primary care clinics as well as from referring physicians or other clinics.
  Healthy controls will be recruited via public announcements and via flyers distributed at a primary care clinic and two universities.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
MR: multi-parameter mapping (MPM) | Once during visit 2 (1-2 weeks after visit 1)
MR: quantitative susceptibility mapping (QSM) | Once during visit 2 (1-2 weeks after visit 1)
Resting-state fMRI (brain and brainstem/spinal cord) | Once during visit 2 (1-2 weeks after visit 1)
MR: whole-brain structural scans | Once during visit 2 (1-2 weeks after visit 1)
MR: routine clinical scans | Once during visit 2 (1-2 weeks after visit 1)
MR spectrosocpy | Once during visit 2 (1-2 weeks after visit 1)
MR: diffusion imaging | Once during visit 2 (1-2 weeks after visit 1)
MR: axial T2*w sequence | Once during visit 2 (1-2 weeks after visit 1)
Task-fMRI | Once during visit 2 (1-2 weeks after visit 1)

SECONDARY OUTCOMES:
Migraine patients: number of migraine attacks, intensity of migraine attacks (intensity 0 - 10), duration, accompanying symptoms, Migraine diary | Once during visit 1 (1-2 weeks prior to visit 2)
Migraine patients: Headache-attributed restriction, disability, social handicap and impaired participation (HARDSHIP) questionnaire | Once during visit 1 (1-2 weeks prior to visit 2)
  Modified questionnaire including personal and socio-demographic, diagnostic questions related to migraine, and enquiry into headache-related burden without strict scale
Migraine/ epilepsy/ visual snow syndrome patients: recording of possible other headache disorders and medication overuse | Once during visit 1 (1-2 weeks prior to visit 2)
HADS questionnaire (Hospital anxiety and depression scale) | Once during visit 1 (1-2 weeks prior to visit 2) for patients and once for healthy participants at MRI visit (1-2 weeks after inclusion into study)
  0-42, higher score > higher probability of anxiety/ depression
Acute medication | Once during visit 1 for patients (1-2 weeks prior to visit 2) and once for healthy participants at MRI visit (1-2 weeks after inclusion into study)
Epilepsy patients: diagnosis and classification according to ILAE | Once during visit 1 (1-2 weeks prior to visit 2)
Epilepsy patients: current anticonvulsant medication | Once during visit 1 (1-2 weeks prior to visit 2)
Epilepsy patients: seizure frequency | Once during visit 1 (1-2 weeks prior to visit 2)
Epilepsy patients: analysis of previous EEG examinations with determination of the epileptic focus (hemisphere, localization) | Once during visit 1 (1-2 weeks prior to visit 2)
Epilepsy patients: analysis of previous EEG examinations with qualitative assessment of the EEG to determine the type of epilepsy-specific abnormalities | Once during visit 1 (1-2 weeks prior to visit 2)
Migraine patients: documentation of previous therapy attempts | Once during visit 1 (1-2 weeks prior to visit 2)
  Which type of therapy (medication, behavioral therapy or neuromodulation)
Epilepsy patients: documentation previous therapy attempts | Once during visit 1 (1-2 weeks prior to visit 2)
  Which type of therapy (medication, surgical intervention or neurostimulation)
Visual snow syndrome: Puledda Questionnaire | Once during visit 2 (1-2 weeks after visit 1)
  The higher the score, the higher the impact of visual snow
Migraine: Dizziness Handicap Inventory (DHI) | Once during visit 2 (1-2 weeks after visit 1)
  Score from 0-100, the higher the score, the higher the vertigo impact

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr. med. Dr. rer. nat., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Klinik Lengg, Zurich
  - University Hospital Zurich, Zurich